CLINICAL TRIAL: NCT07102784
Title: Adapting the Social Cognition and Interaction Training (SCIT) for Early Intervention Psychosis. A Preliminary Qualitative Study.
Brief Title: Adapting a Socio-cognitive Intervention to Early Psychosis Services
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 1075
Record Dates: First submitted 2025-07-30; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Psychoses
Keywords: social cognition; intervention; early onset psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Social cognition (SC) is a broad term used to describe abilities we use to process/interpret emotional cues, others' and own thoughts/feelings. People experiencing psychosis may find dealing with social situations, and interaction with others challenging. Indeed, it is known that SC is impaired in psychosis and this has an impact on social life, ability to live independently, maintain social relationship, and work. Despite the importance of SC in everyday life of people experiencing psychosis there is not a treatment targeting this problem.

The Social Cognition and Interaction Training (SCIT) is a 20-session group intervention developed in the U.S. to help people with psychosis improve their social cognitive skills. More research is needed because SCIT can offer advantages for patients and services in the NHS.

This project aims to prepare some preliminary information for developing a larger study about adapting an adapted version of the SCIT in early psychosis services in SLaM. This adapted version could be shorter or modified on its content.

The goal of this project is to gather information from mental health clinicians (e.g., psychologists) to have their opinions on the SCIT and how/if that can be adapted to early intervention services for psychosis. Interviews will be used to obtain this information. Results from this study will be to develop a larger study involving service users and testing the modified version of the SCIT.

ELIGIBILITY:
Inclusion Criteria:

1. Be either a clinical psychologist, an assistant psychologist, or a trainee clinical psychologist.
2. Have a clinical experience of working with psychosis patients of a minimum of 1 year.
3. Currently working in any of the at-risk mental state for psychosis (through the OASIS service) across any of the four boroughs of the SLaM NHS Foundation Trust: (Southwark, Lambeth, Lewisham and Croydon), and/or in any early intervention (EI) for psychosis services (the Lambeth Early Onset (LEO) service, Southwark EI (STEP), Lewisham EI (LEIS), Croydon EI (COAST).

Exclusion Criteria:

1. Having less than 1 year of clinical working experience with patients suffering from psychosis.
2. Not being employed in any of psychosis services in SLaM NHS Foundation Trust.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinicians delivering psychological intervention to patients experiencing psychosis.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The main outcome of this study is a draft adaptation of the Social Cognition and Interaction Training for Early Intervention Psychosis services. | From August to December 2025